CLINICAL TRIAL: NCT05120583
Title: Incorporation of Pilates-based Core Strengthening Exercises Into the Rehabilitation Protocol for Adolescents With Patellofemoral Pain Syndrome: a Randomized Clinical Trial
Brief Title: Pilates-based Core Strengthening on Patellofemoral Pain Syndrome
Acronym: Pilates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other); Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, College of Medical Rehabilitation, Qassim University, Saudi Arabia, Qassim, Buraidah. Consultant Physical Therapist, El-Sahel Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Cairo, Egypt., Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/20/0049
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; Pilates exercises; functional status
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Patients in the study group received Pilates exercises (25 minutes/ session). There are different types of equipment to be used in Pilates exercises to achieve different purposes; mat, Pilates band or elastic bands, and Pilate's ball were used.
  Interventions: Other: Pilates exercises
- control group (Experimental): Participants in control group received the traditional physical therapy program program (60 minutes/session, three sessions /week for three months).
  Interventions: Other: Traditional physical therapy program

INTERVENTIONS:
Other: Pilates exercises — Side kick internal/ external rotation with Pilate's band
  Other Names: Pilates band
  Arms: study group
Other: Traditional physical therapy program — strength, flexibility
  Other Names: strengthening exercises
  Arms: control group

SUMMARY:
Patellofemoral pain syndrome (PFPS) is one of the most common musculoskeletal pain conditions that tend to become a chronic problem. PFPS is common among young adolescents, particularly in physically active individuals aged 12 to 17 years old with more prevalence among females, as it affects females 1.5 - 3 times when compared to males.

DETAILED DESCRIPTION:
Adolescents with PFPS usually complain of retro-patellar pain (behind the kneecap) or peripatellar pain (around the kneecap) and crepitation in the knee joint, and also there is discomfort while sitting with a flexed knee for a long time. Symptoms are usually exacerbated by activities that increase the load on patellofemoral joints such as weight-bearing activities, squatting, walking up or downstairs, and running.

PFPS takes place whenever the muscles around the knee fail to keep the kneecap properly aligned, leading to abnormal lateral tracking of the patella.Overuse such as running and jumping sports, the trauma of kneecaps such as fracture, dislocation, or knee surgery may also predispose to PFPS.

ELIGIBILITY:
Inclusion Criteria:

* Pain felt anterior to knee joint.
* Pain felt retro-patellar.
* Pain felt during rest and increased with activities like prolonged sitting, squatting, running, and stair climbing.
* Insidious onset lasting for more than 6 weeks.
* Without any traumatic incidence.
* Not participating in a physical therapy program for the past three months.

Exclusion Criteria:

* If they had a meniscal tear.
* Cruciate/collateral ligaments involvement.
* Knee osteoarthritis.
* Rheumatoid arthritis.
* A history of knee or hip surgery.
* Patellar dislocation/subluxation.
* Traction apophysitis encompassing the patellofemoral complex.
* Any pathology in the patellar tendon.
* Spinal referred pain.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Pain assessment | at baseline
  assessed by using a visual analog scale, 10-cm VAS scale, with 0 indicating no pain and 10 for worst pain sensation
Pain assessment | after 12 weeks
  assessed by using a visual analog scale,10-cm VAS scale, with 0 indicating no pain and 10 for worst pain sensation
Muscle strength assessment | at baseline
  assessed using a calibrated handheld dynamometer
Muscle strength assessment | after 12 weeks
  assessed using a calibrated handheld dynamometer

SECONDARY OUTCOMES:
Functional status | at baseline
  evaluated using the Arabic version of the Anterior Knee pain Questionnaire, The score ranges from 0 to 100, with 0 indicating complete functional limitation and 100 indicating no pain and no functional limitation.
Functional status | after 12 weeks
  evaluated using the Arabic version of the Anterior Knee pain Questionnaire, The score ranges from 0 to 100, with 0 indicating complete functional limitation and 100 indicating no pain and no functional limitation.
health-related quality of life | at baseline
  assessed by using the self-report Pediatric Quality of Life Inventory, it includes 23 items distributed among 4 domains [physical (8 items), emotional (5 items), social (5 items), and school functions (3 items)]. Each item is rated on a 5- points scale (0 means never, and 4 means almost always). Items are transformed linearly to 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, and 4 = 0).
health-related quality of life | after 12 weeks
  assessed by using the self-report Pediatric Quality of Life Inventory, it includes 23 items distributed among 4 domains [physical (8 items), emotional (5 items), social (5 items), and school functions (3 items)]. Each item is rated on a 5- points scale (0 means never, and 4 means almost always). Items are transformed linearly to 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, and 4 = 0).

CONTACTS AND LOCATIONS:
Overall Officials: Alshimaa Azab, PhD, Study Director — Cairo University
Locations (1):
- Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Park SK, Stefanyshyn DJ. Greater Q angle may not be a risk factor of patellofemoral pain syndrome. Clin Biomech (Bristol). 2011 May;26(4):392-6. doi: 10.1016/j.clinbiomech.2010.11.015. Epub 2010 Dec 21. PMID 21177007
- [Background] Rabelo ND, Lima B, Reis AC, Bley AS, Yi LC, Fukuda TY, Costa LO, Lucareli PR. Neuromuscular training and muscle strengthening in patients with patellofemoral pain syndrome: a protocol of randomized controlled trial. BMC Musculoskelet Disord. 2014 May 16;15:157. doi: 10.1186/1471-2474-15-157. PMID 24884455
- [Result] Van Der Heijden RA, Lankhorst NE, Van Linschoten R, Bierma-Zeinstra SM, Van Middelkoop M. Exercise for treating patellofemoral pain syndrome: an abridged version of Cochrane systematic review. Eur J Phys Rehabil Med. 2016 Feb;52(1):110-33. Epub 2015 Jul 9. PMID 26158920